CLINICAL TRIAL: NCT06127459
Title: Virtual Reality in Rehabilitation of Executive Functions in Children (VREALFUN)
Brief Title: Virtual Reality in Rehabilitation of Executive Functions in Children With Mild or Moderate Traumatic Brain Injury
Acronym: VREALFUN-TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merja Nikula (Other)
Collaborators: University of Oulu (Other); Aalto University (Other); University of Helsinki (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Merja Nikula, Principal investigator, Oulu University Hospital
Organization: Oulu University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206/ 2021
Record Dates: First submitted 2023-09-28; First posted 2023-11-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Attention; Executive Function; Virtual Reality; Child
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental Guidance+Virtual Reality Game (Experimental)
  Interventions: Behavioral: Parental Guidance; Behavioral: Virtual Reality Game
- Control Group (No Intervention): This group implement the rehabilitation plan drawn up in specialized medical care (treatment as usual).

INTERVENTIONS:
Behavioral: Parental Guidance — Parents get guidance for children's positive behaviour support by using parts of Self-Help Program on the MentalHub.fi (in Finnish: Mielenterveystalo.fi) website regarding children's challenging behaviour (in Finnish: Lasten haastavan käytöksen omahoito-ohjelma).
  Other Names: Self-Help Program of children's challenging behaviour ( Program name in Finnish: Lasten haastavan käytöksen omahoito-ohjelma).
  Arms: Parental Guidance+Virtual Reality Game
Behavioral: Virtual Reality Game — Virtual reality game for rehabilitation of attention, activity control and executive functions by using the virtual environment that corresponds to the typical everyday situations at home.
  Arms: Parental Guidance+Virtual Reality Game

SUMMARY:
Traumatic brain injury (TBI) causes lifelong disability. Children with TBI often have difficulties in attention regulation and executive functions affecting their daily living. Need for rehabilitation is often long-lasting and there is an increasing demand for timely, cost-effective, and feasible rehabilitation methods, where the training is targeted to support daily life functional capacity. The use of Virtual Reality (VR) in the rehabilitation of children with attention and executive function deficits offers opportunities to practice skills required in everyday life in environments emulating real-life situations.

The aim of this research project is to develop a novel effective VR rehabilitation method for children with deficits in attention, activity control, and executive functions by using a virtual environment that corresponds to typical everyday life. In this randomized control study, VR glasses are used to present the tasks, and the levels of difficulty are adjusted according to the child's progress.

The researchers expect that; 1) Intensive training improves the attention regulation, activity control skills, and executive functions of the children in the intervention group 2)Training of executive skills with motivating tasks in a virtual environment that is built to meet challenging everyday situations transfers to the child's everyday life, 3)The duration of the training effect does not depend on the success of the VR training itself, but on how well the child adopts new strategies that make everyday life easier and how the parent is able to support the child's positive behaviour in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate traumatic brain injury (ICD-10: S06.0-S06.6 and S06.8-S06.9 and criteria defined in the Current Care Recommendation, 2021) and
* The challenges of attention and executive function identified in the assessment of a neuropsychologist/experienced psychologist and
* Age 8-12 years and
* Finnish as a native language

Exclusion Criteria:

* Sensitivity to flashing light,
* Epilepsy (ICD-10 G40),
* Mental retardation (ICD-10 F70-F79),
* Pervasive developmental disorders (ICD-10 F84),
* Inflammatory diseases of the central nervous system (ICD-10 G00-G09),
* Severe cerebral palsy syndrome (ICD-10 G80, GMFCS 4-5, MACS 3-5),
* Brain tumour, and
* Multiple pregnancy

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Epeli (Executive Performance in Everyday LIving) task | Baseline, 4-6 weeks, 6 months and 12 months.
  A virtual reality task for attention, executive function, and prospective memory. Change in total score, task efficacy, navigation efficacy, controller motion, and total action.
ADHD-rating scale IV (ADHD-RS) (parent report) | Baseline, 4-6 weeks, 6 months and 12 months.
  The ADHD-RS (parent report) is an assessment of a child's ADHD symptoms with 18 items based on the child's behaviour over the past 6 months. 4-point Likert scale. The total score ranges 0-54, scores in inattention subscale and hyperactivity/impulsivity subscale range 0-27. Change in the total score, inattention subscale score, and hyperactivity/impulsivity subscale score on a parent-rated ADHD-RS. A lower score means a better outcome.
Epeli Questionnaire (parent report) | Baseline, 4-6 weeks, 6 months and 12 months.
  An assessment of a child's functional ability and the amount of positive feedback given by the parent to the child over the past 4 weeks. 5-point Likert scale. 2 subscales: Functional ability subscale where score ranges 4-20, and Positive feedback subscale where score ranges 4-20. Change in Functional ability subscale score and Positive feedback subscale score on parent-rated Epeli- questionnaire. A higher score means a better outcome.
Epeli Questionnaire (child report) | Baseline, 4-6 weeks, 6 months and 12 months.
  An assessment of a child's functional ability and the amount of positive feedback given by the parent to the child over the past 4 weeks. 5-point Likert scale. 2 subscales: Functional ability subscale where score ranges 4-20, and Positive feedback subscale where score ranges 4-20. Change in Functional ability subscale score and Positive feedback subscale score on child-rated Epeli- questionnaire. A higher score means a better outcome.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF-2) (parent form) | Baseline, 4-6 weeks, 6 months and 12 months.
  A measure of executive functions of children and adolescents in natural settings containing 63 items rated by the parent. 3-point Likert scale. Change in Global Executive Composite score, Behavior regulation score, Emotion regulation score, and Cognitive regulation score on parent-rated BRIEF-2. In case the data in the Behavior regulation, Emotion regulation, and Cognitive regulation subscales are not too strongly correlated (r<0.7) and there will be a significant effect of the intervention on the BRIEF-2 Global Executive Composite score, we will use the subscales to conduct a post hoc analysis examining which domains of executive functions are affected. A higher score means a worse outcome.
Behavior Rating Inventory of Executive Function (BRIEF-2) (teacher form) | Baseline, 4-6 weeks, 6 months and 12 months.
  A measure of executive functions of children and adolescents in natural settings containing 63 items rated by the teacher. 3-point Likert scale. Change in Global Executive Composite score, Behavior regulation score, Emotion regulation score, and Cognitive regulation score on teacher-rated BRIEF-2. In case the data in the Behavior regulation, Emotion regulation, and Cognitive regulation subscales are not too strongly correlated (r<0.7) and there will be a significant effect of the intervention on the BRIEF-2 Global Executive Composite score, we will use the subscales to conduct a post hoc analysis examining which domains of executive functions are affected. A higher score means a worse outcome.
Concentration questionnaire (in Finnish: Keskittymiskysely) | Baseline, 4-6 weeks, 6 months and 12 months.
  An assessment of attention and executive function difficulties in school-aged children with 55 items. 3-point Likert Scale, Total score range 0-110. Change in Total score, Distractibility score (range 0-8), sum of Impulsivity and Motor hyperactivity subscales scores (range 0-32), sum of Directing, Sustaining and Shifting Attention subscales scores (range 0-30), and sum of Initiative, Planning, Execution and Evaluation of Action subscales scores (range 0-40) on teacher-rated Concentration questionnaire. In case the data in the Distractibility subscale, Impulsivity and Motor hyperactivity subscales, Attention subscales and Executive subscales are not too strongly correlated (r<0.7) and there will be a significant effect of the intervention on Concentration questionnaire Total score, we will use the subscales to conduct a post hoc analysis examining which domains of executive functions are affected. A higher score implies a worse outcome.
Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents Revised Version ( KINDL-R) (parent version) | Baseline, 4-6 weeks, 6 months and 12 months.
  An assessment of Health-Related Quality of Life in children and adolescents with 24 items. 5-point Likert scale. Change in Total score on parent-rated questionnaire. A higher score means a better outcome.
9. Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents Revised Version (KINDL-R) (self-report version) | Baseline, 4-6 weeks, 6 months and 12 months.
  An assessment of Health-Related Quality of Life in children and adolescents with 24 items. 5-point Likert scale. Change in Total score on child-rated questionnaire. A higher score means a better outcome.
N-back test | Baseline, 4-6 weeks, 6 months and 12 months.
  A test for a working memory. Change in 2-back and 1-back hitrate and reaction time.
The Conners Continuous Performance Test 3rd Edition (Conners CPT3) | Baseline, 4-6 weeks, 6 months and 12 months.
  A computerized attention task validated in individuals aged 8 years and older. Change in scores on Conners Continuous Performance Test (CPT-3).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Uusimaa, MD, PhD, Study Chair — Oulu University Hospital; Merja Nikula, M.Psych., Principal Investigator — Oulu University Hospital; Mirjami Mäntymaa, MD, PhD, Study Director — Oulu University Hospital; Juha Salmitaival, PhD, Study Director — Aalto University, Finland; Elias Ollikainen, B.M., Principal Investigator — University of Oulu, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland